CLINICAL TRIAL: NCT00571129
Title: Recovery After Endoscopic Dacryocystorhinostomy
Brief Title: Endoscopic Dacryocystorhinostomy Prospective Research
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Juha Seppa, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5551812; 255104 (Other: Kuopio University Hospital)
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Lacrimal Duct Obstruction
Keywords: Primary,silicone tube,revision,mitomycin C,endoscopic DCR
MeSH Terms: conditions — Lacrimal Duct Obstruction | interventions — Mitomycin

STUDY DESIGN:
Intervention Model Description: DCR with/ without tubes Revision DCR with/ without mitomycin
Oversight: Data Monitoring Committee: No

ARMS (2):
- with tubes or mitomycin (Active Comparator): After DCR bicanalicular tubes were inserted After re-DCR mitomycin in cottonpads were placed into rhinostoma for 5 minutes
  Interventions: Procedure: DCR with no tubes or mitomycin
- without tubes or mitomycin (Active Comparator): After DCR no tubes were inserted After re-DCR no mitomycin was used
  Interventions: Procedure: DCR with no tubes or mitomycin

INTERVENTIONS:
Procedure: DCR with no tubes or mitomycin — The patients were randomized into the two study groups, either with or without the insertion of a bicanalicular silicone tube after primary DCR.
  In revision group patients were randomized into the two groups,ether with or without application of mitomycin "C" after DCR
  Other Names: DCR with tubes or mitomycin

SUMMARY:
Endoscopic dacryocystorhinostomy (EN-DCR) is an effective procedure when treating saccal and postsaccal obstructions of the nasolacrimal pathway. The benefit of silicone tubing after DCR is still controversial. We conducted a prospective, randomized study in order to evaluate 1) the necessity of bicanalicular silicone tubes after primary EN-DCR, 2) efficacy of the perioperative Mitomycin C for the prevention of adheesion and re-stenosis of rhinostomy site in revision EN-DCR, 3) the subjective symptoms and QoL changes before and after DCR-operation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age > 18), ASAI-III, and were scheduled for primary or revision lacrimal pathway surgery due to recurrent or chronic watering eyes or conjunctival discharge.
* Patients were excluded if they had previous nasolacrimal surgery, malignancy in the paranasal sinuses, nasal cavity, or lacrimal pathway, presaccal obstruction, pregnancy or lactation, or mental disability.

Exclusion Criteria:

* Malignancy in the paranasal sinuses, nasal cavity, or lacrimal pathway, presaccal obstruction, pregnancy or lactation, or mental disability.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-09 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The success rate after primary DCR with and without silicone tubes. The success rate after revisio DCR with and without Mitomycin C. | 5 years

SECONDARY OUTCOMES:
The EN-DCR operation influence on the patients subjective symptoms and QoL before and after operation. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Juha Seppä, MD,PhD, Study Chair — Kuopio University Hospital, Otorhinolaryngology
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

REFERENCES:
- [Background] Penttila E, Hyttinen JM, Hytti M, Kauppinen A, Smirnov G, Tuomilehto H, Seppa J, Nuutinen J, Kaarniranta K. Upregulation of inflammatory genes in the nasal mucosa of patients undergoing endonasal dacryocystorhinostomy. Clin Ophthalmol. 2014 Apr 25;8:799-805. doi: 10.2147/OPTH.S50195. eCollection 2014. PMID 24851037